CLINICAL TRIAL: NCT02506803
Title: Phase I Study of Neoadjuvant Chemotherapy of Gemcitabine Plus Nab-paclitaxel for Patients With Borderline Resectable Pancreatic Cancer.
Brief Title: Phase I Study of Neoadjuvant Chemotherapy for Patients With Borderline Resectable Pancreatic Cancer.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wakayama Medical University (Other)
Responsible Party: Principal Investigator, Hiroki Yamaue, Dean & Professor of the second department of surgery, Wakayama Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAC-GEMABR
Record Dates: First submitted 2015-07-22; First posted 2015-07-23 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NAC-GEMABR (Experimental): Neoadjuvant chemotherapy 2 courses of NAC-GEMABR for subsequent 10 patients.
  Interventions: Drug: NAC-GEMABR

INTERVENTIONS:
Drug: NAC-GEMABR — NAC-GEMABR regimen includes gemcitabine 1000mg/m2 plus nab-paclitaxel 125mg/m2 3 times weekly 1week rest.
  Other Names: Gemcitabine, nab-paclitaxel

SUMMARY:
Gemcitabine plus nub-paclitaxel (GEMABR) regimen was recently presented at an international oncology meeting and represents a new standard regimen in the treatment of metastatic pancreatic cancer. Therefore, it was decided to consider the balance of safety and efficacy as a preoperative chemotherapy, the investigators use the NAC-GEMABR regimen includes only two cycles (three times weekly and one week rest) of GEMABR regimen.

DETAILED DESCRIPTION:
Gemcitabine plus nub-paclitaxel (GEMABR) regimen was recently presented at an international oncology meeting and represents a new standard regimen in the treatment of metastatic pancreatic cancer. GEMABR is one of the high response rate treatment regimen, the investigators considered as a promising treatment as neoadjuvant chemotherapy . On the other hand , incidences of grade 3 or 4 neutropenia , febrile neutropenia and peripheral neuropathy were significantly higher in the g group compared with gemcitabine group. Therefore, it was decided to consider the balance of safety and efficacy as a preoperative chemotherapy, the investigators use the NAC-GEMABR regimen includes only two cycles (three times weekly and one week rest) of GEMABR regimen. The investigators also evaluate the optimal treatment schedule of NAC-GEMABR therapy as neoadjuvant chemotherapy, optimal duration between surgery and chemotherapy, R0 resection rate, and resection rate for borderline resectable pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven invasive pancreatic ductal carcinoma
* Cases that meet the definition of borderline resectable pancreatic cancer 1) or 2)

  1. Definition of a borderline resectable pancreatic cancer is filledin NCCN guideline version 1.2014 pancreatic adenocarcinoma
  2. Patients indicated distal pancreatectomy with en bloc celiac axis resection
* PS (ECOG) 0-1
* ≧20 years old and < 80 years old
* First line treatment
* The following criteria must be satisfied in laboratory tests within 14 days of registration White blood cell count ≦12,000/mm3 Neutrophil count ≧1,500/mm3 Platelet count ≧100,000mm3 Total bilirubin <2.0mg/dL Serum Creatinine ≦upper limits of normal(ULN) AST, ALT≦2.5×ULN Albumin≧3.0g/dL Hemoglobin≧9.0g/dL
* Written informed consent to participate in this study

Exclusion Criteria:

* Severe drug hypersensitivity
* Multiple primary cancers within 5 years
* Severe infection
* With grade2 or more severe peripheral neuropathy
* With intestinal paralysys, ileus
* Interstitial pneumonia or pulmonary
* With uncontrollable pleural effusion or ascites
* Receiving atazanavir sulfate
* With uncontrollable diabetes
* With uncontrollable heart failure, angina, hypertension, arrhythmia
* With severe psychological symptoms
* With watery diarrhea
* Pregnant or lactating women, or women with known or suspected pregnancy
* Inappropriate patients for entry on this study in the judgment of the investigator

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with toxicity of NAC-GEMABR therapy as neoadjuvant chemotherapy for borderline resectable pancreatic cancer. | Up to 30 weeks.
  Toxicities will be assessed according to Common Terminology Criteria for Adverse Events (CTCAE) 4.0.

SECONDARY OUTCOMES:
The resection rate of NAC-GEMABR therapy as neoadjuvant chemothterapy for borderline resectable pancreatic cancer. | Up to 24 weeks
The R0 resection rate of NAC-GEMABR therapy as neoadjuvant chemotherapy for borderline resectable pancreatic cancer. | Up to 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hiroki Yamaue, M.D., PhD, Principal Investigator — Wakayama Medical University
Locations (1):
- Wakayama Medical University, Wakayama, Japan

REFERENCES:
- [Derived] Okada KI, Hirono S, Kawai M, Miyazawa M, Shimizu A, Kitahata Y, Ueno M, Hayami S, Yamaue H. Phase I Study of Nab-Paclitaxel plus Gemcitabine as Neoadjuvant Therapy for Borderline Resectable Pancreatic Cancer. Anticancer Res. 2017 Feb;37(2):853-858. doi: 10.21873/anticanres.11389. PMID 28179342